CLINICAL TRIAL: NCT02773745
Title: The Effects of Aquatic Prehabilitation in Knee OA Patients on Knee Arthroplasty Outcomes
Brief Title: Prehabilitation Using Aquatic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00032580
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participant will receive standard of care and a brochure on healthy eating.
- Aquatic Prehabilitation Group (Active Comparator): The prehabilitation group will undergo 6-8 weeks of individualized aquatic exercise in a heated pool (60 min/session, 3 times per week). Aquatic equipment maybe used to challenge balance and trunk stabilization.
  Interventions: Behavioral: Aquatic Prehab

INTERVENTIONS:
Behavioral: Aquatic Prehab — Pool therapy
  Arms: Aquatic Prehabilitation Group

SUMMARY:
With aging population, total knee arthroplasty is performed with increasing frequency. Although the surgery is successful in general, significant number of patients suffers persistent pain and disability. Traditional risk assessment tool have been focused on single organ systems. Our investigators have found that mobility, assessed by the Mobility Assessment Tool short form (MAT-sf), is a simple and accurate method to predict postoperative outcome, including length of stay, postoperative complications, and nursing home placement for older patients. Prehabilitation is the process of enhancing a person's functional capacity to withstand an incoming stressor. Although multiple studies have tested prehabilitation before joint replacement surgery, results have been mixed. The investigators hypothesize that patients with limited mobility are most likely to benefit from prehabilitation. The investigators plan to use individualized aquatic exercise as a prehabilitation tool to enhance compliance; the resistance of water strengthen muscle and increasing energy expenditure; the buoyancy of water provides environment where the joints are not weight bearing. The aims of the study are: 1) To evaluate the feasibility of prehabilitation using 6-8 weeks of aquatic exercise in 40 geriatric patients who are scheduled for total knee arthroplasty for osteoarthritis; 2) To examine the effects of 6-8 weeks of aquatic exercise on mobility, pain, stiffness, physical function, cognitive function and depression; inflammatory markers and 3) To estimate the effect of prehabilitation on postoperative outcomes. The investigators plan to enroll 40 patients age >50, who are scheduled for elective primary total knee replacement. Investigators will screen patients in the Preoperative Assessment Clinic and enroll patients who have decreased mobility, measured by MAT-sf. Patients will be randomized into either a prehabilitation group or a usual care group. All the participants will undergo extensive assessment on their pain, stiffness, and physical function, depression, balance and cognitive function using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the expanded Short Physical Performance Battery (eSPPB), and Montreal Cognitive Assessment (MoCA). Serum inflammatory markers will be assessed at the baseline. The prehabilitation group will undergo 6-8 weeks of individualized aquatic exercise in a heated pool (60 min/session, 3 times per week). Aquatic equipment maybe used to challenge balance and trunk stabilization. All participants will be reassessed immediately before surgery and 4 weeks after the surgery using WOMAC, eSPPB, MoCA and MAT-sf. Serum inflammatory markers and body composition will be reassessed at the same time points. The primary outcome of interest is will be postoperative complications, length of stay, Intensive Care Unit length of stay, and institutionalization. If successful, investigators will have sound pilot data for several critical health outcomes with which to support an external proposal for a larger-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Age > 50
* Willingness to exercise in a pool 3 times a week
* MAT-Sf score ≤ 58 for men and ≤ 50 for women
* Participant is scheduled for primary total knee replacement surgery due to OA >4 weeks from expected BV visit
* Not involved in any other behavioral, exercise or investigational drug intervention study

Exclusion Criteria:

* Impaired cognitive function (MoCA <21)
* Undergoing knee replacement surgery for indications other than OA
* Undergoing bilateral knee replacements
* Major deficits in hearing or vision
* Currently exercising more than 3 times per week
* Severe depression (GDS-sf ≥ 12)
* Contraindications to the pool: open wounds/ incontinence/history of seizures in last year

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Change in physical function using the MAT-sf | 4-6 weeks after surgery
  Change in MAT-sf score from baseline (prior to surgery) to follow up (4-6 weeks after surgery)
Change in physical function using the eSPPB | 4-6 weeks after surgery
  Change in eSPPB score from baseline (prior to surgery) to follow up (4-6 weeks after surgery)
Change in physical function using the Postural Sway Force Plate | 4-6 weeks after surgery
  Change in postural sway score from baseline (prior to surgery) to follow up (4-6 weeks after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Sunghye Kim, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Clinical Research Unit, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No